CLINICAL TRIAL: NCT07114432
Title: An Exploratory Clinical Study on the Safety and Efficacy of BCMA/CD19 Allogeneic CAR-T Cell Injection in Newly Diagnosed High-Risk Cytogenetic Multiple Myeloma Patients Ineligible or Unwilling to Undergo ASCT
Brief Title: RN1201 Injection in Newly Diagnosed High-Risk Cytogenetic Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Allorunning Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NDHR
Record Dates: First submitted 2025-07-28; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Newly Diagnosed High-Risk Cytogenetic Multiple Myeloma Patients Ineligible or Unwilling to Undergo ASCT; Newly Diagnosed Multiple Myeloma (NDMM)
Keywords: Newly Diagnosed; High-Risk Cytogenetic; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic CAR-T cell therapy (Experimental): Newly Diagnosed High-Risk Cytogenetic Multiple Myeloma Patients Ineligible or Unwilling to Undergo ASCT are treated with allogeneic CAR-T cell therapy
  Interventions: Drug: BCMA/CD19-targeted allogeneic CAR-T

INTERVENTIONS:
Drug: BCMA/CD19-targeted allogeneic CAR-T — Lymphodepletion chemotherapy followed by allogeneic CAR-T cell (RN1201) infusion
  Other Names: RN1201

SUMMARY:
This is a single-arm, dose-escalation exploratory study evaluating the safety and efficacy of RN1201, a BCMA/CD19-targeted allogeneic CAR-T cell therapy, in patients with newly diagnosed cytogenetically high-risk multiple myeloma who are ineligible or unwilling to undergo autologous stem cell transplantation (ASCT). Patients will receive lymphodepletion followed by a single infusion of RN1201 across four dose levels. Primary endpoints include incidence and severity of treatment-emergent adverse events. Secondary endpoints assess response rate and minimal residual disease (MRD) status.

DETAILED DESCRIPTION:
This is a Phase 1, single-arm, dose-escalation exploratory study to evaluate the safety, feasibility, and preliminary efficacy of RN1201, a BCMA/CD19-targeted allogeneic CAR-T cell therapy, in patients with newly diagnosed high-risk cytogenetic multiple myeloma (MM) who are ineligible or unwilling to undergo autologous stem cell transplantation (ASCT). Patients will receive lymphodepletion chemotherapy followed by a single infusion of RN1201 cells, across four dose levels. The primary endpoint will assess the incidence and severity of treatment-emergent adverse events (TEAEs), while secondary endpoints will evaluate the objective response rate (ORR), complete response (CR), minimal residual disease (MRD) status, and pharmacokinetics (PK) and pharmacodynamics (PD) of RN1201.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for this trial only if all of the following criteria are met:

  1. Is willing and able to provide a written informed consent form before any trial-related activities are performed.
  2. Must have a diagnosis of Multiple Myeloma (MM) according to the World Health Organization (WHO) 2017 revised criteria.

     * Must be diagnosed with active MM according to the International Multiple Myeloma Working Group (IMWG) criteria.
     * Must meet the definition of genetic high-risk MM as per the "2024 Chinese Expert Consensus on the Diagnosis and Treatment of High-Risk Multiple Myeloma", defined as having one or more of the following high-risk cytogenetic abnormalities (HRCA) confirmed by FISH or mitotic karyotype analysis:

     del(17p) TP53 mutation t(4;14) t(14;16) t(14;20) 1q21 gain/amplification (defined as copy number ≥ 4) Del 1p Note: 1q21 amplification alone does not define cytogenetic high risk.
  3. Must have a documented MM type that is B-cell maturation antigen (BCMA) positive and/or CD19 positive, confirmed at screening or from prior medical records.
  4. Age ≥ 18 years, male or female.
  5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 at enrollment.
  6. Has a life expectancy of ≥ 12 weeks.
  7. Meets the following prior therapy requirements:

     * Is currently receiving or has received an induction therapy regimen containing at least a proteasome inhibitor, an immunomodulatory agent, or a monoclonal antibody as a backbone therapy.
     * Has not received more than 4 cycles of induction therapy at the time of enrollment.
     * Has had an effective response to induction therapy without evidence of disease progression per IMWG criteria.
     * Prior radiotherapy is permitted before enrollment.
     * Is scheduled to initiate maintenance and/or consolidation therapy 3 months after cell reinfusion, following successful enrollment.
  8. Must have measurable disease to assess Progression-Free Survival (PFS). Measurable disease is defined by at least one of the following criteria:

     * Serum M-protein (M-spike) ≥ 0.5 g/dL.
     * 24-hour urine M-protein (M-spike) ≥ 200 mg.
     * Abnormal serum free light chain (FLC) ratio with an involved FLC level ≥ 50 mg/L.
     * For IgA MM: total serum IgA level outside the normal range.
     * Note: The presence of measurable disease is not required at enrollment; it can be determined from historical lab data. For instance, a subject who achieved a complete response after induction and has no measurable disease at enrollment is still eligible if they met any of the above criteria after their initial diagnosis.
  9. Adequate organ function as defined by the following laboratory values:

     * Total serum bilirubin < 2 times the upper limit of normal (ULN).
     * Serum creatinine < ULN.
     * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) < 3 times ULN.
  10. Estimated or calculated creatinine clearance (CrCl) ≥ 40 mL/min, via CKD-EPI or Cockcroft-Gault formula.
  11. Diffusing capacity of the lungs for carbon monoxide (DLCO) ≥ 50% of predicted value (corrected or uncorrected for anemia/alveolar volume).
  12. Adequate bone marrow function defined as: Absolute neutrophil count ≥ 0.5×10⁹/L and platelet count ≥ 20×10⁹/L.
  13. ECOG performance status of 0-2.
  14. Left ventricular ejection fraction (LVEF) ≥ 50% with no pericardial effusion.
  15. Must have recovered to ≤ Grade 1 (per CTCAE) from any Serious Adverse Event (SAE) before enrollment.
  16. Able to comply with the study visit schedule and other protocol requirements.

Exclusion Criteria:

* A subject will not be eligible for this trial if any of the following criteria are met:

  1. Known history of allergic reaction, hypersensitivity, intolerance, or contraindication to the BCMA/CD19 allogeneic CAR-T product or any of its excipients, including fludarabine, cyclophosphamide, and tocilizumab.
  2. Diagnosis of plasma cell leukemia.
  3. Presence of non-paraskeletal extramedullary disease.
  4. Relapse after allogeneic hematopoietic stem cell transplantation (allo-HSCT) with active graft-versus-host disease (GVHD) that requires treatment with steroids or immunosuppressive agents.
  5. Presence of a severe, active infection, including:

     * Human Immunodeficiency Virus (HIV) infection (subjects must have a negative HIV 1/2 antibody screen).
     * Hepatitis C Virus (HCV) infection (subjects must have a negative anti-HCV antibody screen).
     * Hepatitis B Virus (HBV) infection (subjects must have a negative HBsAg screen).
  6. History of prior gene therapy or genetically modified cell immunotherapy.
  7. Active autoimmune disease, including connective tissue disease, uveitis, sarcoidosis, inflammatory bowel disease, or multiple sclerosis; or a history of a severe autoimmune disease (as judged by the Principal Investigator) that required long-term immunosuppressive therapy.
  8. Diagnosis of an acquired or congenital immunodeficiency disease.
  9. History of Class III or IV heart failure as defined by the New York Heart Association (NYHA), unstable angina, myocardial infarction within the last 6 months, or sustained (>30 seconds) ventricular arrhythmia.
  10. History of seizure disorder or other central nervous system (CNS) disease; history or current evidence of CNS involvement with MM. Note: CNS screening (e.g., lumbar puncture) is not mandatory unless symptoms are present.
  11. History of other primary malignancies, except for the following:

      * Non-melanoma skin cancer (e.g., basal cell carcinoma) cured by resection.
      * Carcinoma in situ (e.g., cervical, bladder, or breast cancer) that has been cured.
  12. Is pregnant, breastfeeding, or, for female subjects, is planning a pregnancy within 6 months.
  13. Participation in another clinical trial within the last month.
  14. Any condition which, in the opinion of the investigator, would place the subject at increased risk or interfere with the trial results.
  15. Has undergone major surgery within 14 days prior to the first dose of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of dose-limiting toxicities (DLTs) | DLTs: Within 28 days after CAR-T cell infusion
The incidence and severity of treatment-emergent adverse events (TEAEs) | TEAEs: From infusion up to 24 months post-treatment.

SECONDARY OUTCOMES:
Overall effectiveness and duration of efficacy | 4 weeks, 3 months, 6 months, and 12 months
  Overall response rate (ORR) and complete response rate (CR), negative rate of MRD (detected by flow cytometry or NGS)
Pharmacokinetic (PK) of RN1201 | From RN1201 infusion up to 12 months
  Levels of RN1201 CAR-positive T cells in the blood and/or bone marrow
Levels of Peripheral blood M protein | From RN1201 infusion up to 12 months
  Levels of Peripheral blood M protein
Levels of urine M protein | From RN1201 infusion up to 12 months
  Levels of urine M protein
Levels of Peripheral blood cytokine | From RN1201 infusion up to 12 months
  Levels of Peripheral blood cytokine, including IL-2, IL-6, IL-10, TNFa et. al.

CONTACTS AND LOCATIONS:
Overall Officials: Yafei Wang, PhD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (2):
- China (2):
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No
Data sharing can be permitted after approval by the study leader due to patient privacy concerns.